CLINICAL TRIAL: NCT01474876
Title: Multicountry Post-Marketing Observational Study on Maintenance of Effectiveness of Adalimumab in Patients With Ankylosing Spondylitis and Psoriatic Arthritis
Brief Title: Multi-country Post-Marketing Observational Study on Maintenance of Effectiveness of Adalimumab (Humira®) in Patients With Ankylosing Spondylitis and Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-768
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Post-marketing observational study (PMOS) Protocol; Effectiveness of Adalimumab (HUMIRA®); Psoriatic Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis: Participants with a diagnosis of ankylosing spondylitis
- Psoriatic Arthritis: Participants with a diagnosis of psoriatic arthritis

SUMMARY:
This 12-month postmarketing observational study (PMOS) was a prospective, single-arm, multicenter, multi-country study, with follow-up visits at 3, 6, 9, and 12 months after the initial baseline visit. The study was conducted to determine the long-term effectiveness of treatment with adalimumab in routine clinical use in participants with Ankylosing Spondylitis (AS) and Psoriatic Arthritis (PsA) in Central and Eastern European Countries.

DETAILED DESCRIPTION:
Additional study objectives were to evaluate AS and PsA with regard to extra-articular manifestations (EAMs), functional status, the use of concomitant nonsteroidal anti-inflammatory medication, and work productivity impairment. In addition, the Ankylosing Spondylitis Disease Activity Score (ASDAS), a new disease activity index in AS, was measured in parallel with the standard Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score to assess the effectiveness of adalimumab in treating axial symptoms.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled in this Postmarketing observational study PMOS if they fulfill all of the below criteria:

1. Adult patients with diagnosis of Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA).
2. Eligible for adalimumab therapy according to the local product label and prescription/reimbursement guidelines.
3. Have been prescribed adalimumab within a maximum of one (1) month prior to the study enrolment.
4. Have negative result of Tuberculosis (TB) screening test or TB prophylaxis as per local guidelines.
5. Are willing to provide Authorization to the investigator to use and/or disclose personal and/or health data, or to provide Informed Consent if requested by the Local Regulations, before entry into the study.

Exclusion Criteria:

Patients fulfilling below exclusion criteria will not be eligible for this Postmarketing study (PMOS):

1. Meet contraindications for treatment with adalimumab as outlined in the latest version of the local Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a post-marketing observational study (PMOS) where adalimumab is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. Study population will consist of adult aged (>18 years) with Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA) that can be administered adalimumab as per locally approved Summary of Product Characteristics (SmPC) and reimbursement criteria.
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isidro Villanueva Torrecillas, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 566 participants were enrolled, and 11 participants were lost to follow-up after the baseline visit. According to the pre-specified analysis strategy in the statistical analysis plan, these participants were excluded from the full analysis set, which consisted of 555 participants.
Groups:
- Disease State Unknown: For one participant, information regarding the underlying disease was not available
Period: Overall Study
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Disease State Unknown
Started | 403 | 151 | 1
Completed | 337 | 128 | 1
Not Completed | 66 | 23 | 0
Not completed — Adverse Event | 11 | 5 | 0
Not completed — Serious Adverse Event | 2 | 3 | 0
Not completed — Lost to Follow-up | 5 | 4 | 0
Not completed — Investigator's decision | 28 | 6 | 0
Not completed — Patient's request | 19 | 5 | 0
Not completed — Investigator's decision and pt request | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received adalimumab treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis | Disease State Unknown | Total
Number analyzed (Participants) | 403 | 151 | 1 | 555
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.8) | 49.7 (12.1) | 40 (NA) — n=1 participant | 45.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 65 | 0 | 174
  Male | 294 | 86 | 1 | 381

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 50% or More Decrease in Bath Ankylosing Spondylitis Daily Activity Index (BASDAI) Score at 12 Months Relative to Baseline
Description: The BASDAI score was calculated using a questionnaire with 6 questions that the participants completed by marking responses on a 10-centimeter visual analog scale ranging from 0 (none) to 10 (very severe) regarding severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. A positive response was defined as a 50% or more decrease in the BASDAI score at 12 months as compared to baseline.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with active axial symptoms (a baseline value of the BASDAI > 4).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 366 | 52
Percentage of participants | 76.5 [71.8 to 80.8] | 73.1 [59.0 to 84.4]

2. Primary Outcome: Percentage of Participants With a Disease Activity Score 28 (DAS28) Decrease ≥1.2 at 12 Months Relative to Baseline
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with peripheral symptoms (DAS28 > 5.1 at baseline)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 18 | 61
Percentage of participants | 83.3 [58.6 to 96.4] | 83.6 [71.9 to 91.8]

3. Primary Outcome: Percentage of Participants With Active Axial Symptoms in Remission
Description: The Ankylosing Spondylitis Disease Score (ASDAS) tool is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, duration of morning stiffness and peripheral pain/swelling assessed on a visual analogue scale (from 0 to 10 cm) or on a numerical rating scale (from 0 to 10). The laboratory parameter is a measurement of C-reactive protein (mg/L) or erythrocyte sedimentation rate (mm/h). Remission was defined as ASDAS <1.3 at 12 months.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with active axial symptoms (a baseline value of BASDAI > 4)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 361 | 52
Percentage of participants | 34.3 [29.5 to 39.5] | 28.8 [17.1 to 33.1]

4. Secondary Outcome: Mean Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score (in Case of Axial Symptoms) and/or Disease Activity Score/28 Joints (DAS28) (in Case of Peripheral Symptoms) in Participants With Ankylosing Spondylitis
Description: The BASDAI score was calculated using a questionnaire with 6 questions that the participants completed by marking responses on a 10-centimeter visual analog scale ranging from 0 (none) to 10 (very severe) regarding severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. A positive response was defined as a 50% or more decrease in the BASDAI score at 12 months as compared to baseline.
  The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C- reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with ankylosing spondylitis with peripheral symptoms (DAS28 > 5.1 at baseline) and/or active axial symptoms (a baseline value of BASDAI > 4)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 366
Units on a scale
  Mean change in BASDAI score, n=366 | -4.6 (2.3)
  Mean change in DAS28 score, n=18 | -1.9 (1.3)

5. Secondary Outcome: Mean Change in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, and peripheral pain/swelling assessed on a visual analogue scale (from 0 (normal) to 10 (extreme pain or disability) cm) and duration of morning stiffness on a numerical rating scale (from 0 to 10, with 0 being none and 10 representing a duration of 2 hours or longer). The laboratory parameter is a measurement of C-reactive protein (mg/L) (CRP) or erythrocyte sedimentation rate (mm/h) (ESR). Data from five variables (disease activity, back pain, duration of morning stiffness, peripheral pain/swelling, and either CRP or ESR values) are combined to yield a score ranging from 0 to no defined upper limit. Remission is defined as ASDAS score <1.3. Clinically important improvement is defined as a change ≥ 1.1 units, and major improvement is defined as a change ≥ 2.0 units.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with active axial symptoms (a baseline value of BASDAI > 4)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 358 | 51
Units on a scale
  Mean change in ASDAS-CRP, n=299 and 45 | -2.6 (1.2) | -1.9 (1.7)
  Mean change in ASDAS-ESR, n=358 and 51 | -2.3 (1.1) | -1.9 (1.4)

6. Secondary Outcome: Correlation Between Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Ankylosing Spondylitis Disease Activity Score (ASDAS) in Participants With Ankylosing Spondylitis
Description: BASDAI score (ranging from 0 to 10) was calculated using a questionnaire. Participants marked responses on a 10 cm visual analog scale ranging from 0 (none) to 10 (very severe) regarding fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. A positive response was defined as a 50% or more decrease in the BASDAI score at 12 months as compared to baseline. ASDAS is a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, duration of morning stiffness and peripheral pain/swelling assessed on a visual analogue scale (from 0 to 10 cm) or on a numerical rating scale (from 0 to 10). The laboratory parameter is a measurement of C-reactive protein (mg/L) or erythrocyte sedimentation rate (mm/h). Spearman's rank correlation coefficient (CC) was calculated for BASDAI vs. ASDAS(subscript)CRP(subscript) and BASDAI vs. ASDAS(subscript)ESR(subscript ).
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with ankylosing spondylitis and active axial symptoms (a baseline value of BASDAI > 4)
Measure: Number; unit: Correlation coefficient
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 358
Correlation coefficient
  Correlation BASDAI and ASDAS-CRP, n=299 | 0.62
  Correlation BASDAI and ASDAS-ESR, n=358 | 0.71

7. Secondary Outcome: Predictors of Maintained Treatment Response and Remission in Participants With Ankylosing Spondylitis
Description: A mathematical technique called logistic regression was performed to identify factors that could be used to predict maintained treatment response and remission. The following baseline variables were used in the logistic regression analyses: age, gender, disease of interest, result of tuberculosis screening, time since diagnosis and extra-articular manifestations (symptoms and diseases that occur in parts of the body other than joints) at baseline. The BASDAI score at baseline was forced to serve as a predictor in each model.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with ankylosing spondylitis and active axial symptoms (a baseline value of BASDAI > 4)
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 361
Odds Ratio
  Response (Age), n=361 | 0.98 [0.96 to 1.00]
  Response (Enthesitis at V0), n=361 | 2.47 [1.15 to 5.27]
  Response (BASDAI at V0), n=361 | 1.18 [0.98 to 1.42]
  Remission (Age), n=356 | 0.96 [0.95 to 0.98]
  Remission (TB positive at V0), n=356 | 0.57 [0.30 to 1.06]
  Remission (Male gender), n=356 | 1.77 [1.02 to 3.08]
  Remission (BASDAI at V0), n=356 | 0.94 [0.80 to 1.12]
Statistical Analysis 1: Comparison: Ankylosing Spondylitis; Treatment response and participant age; Test type: Superiority or Other; p = 0.0164, Regression, Logistic
Statistical Analysis 2: Comparison: Ankylosing Spondylitis; Treatment response and presence of enthesitis at Visit 0; Test type: Superiority or Other; p = 0.0200, Regression, Logistic
Statistical Analysis 3: Comparison: Ankylosing Spondylitis; Treatment response and BASDAI score at Visit 0; Test type: Superiority or Other; p = 0.0867, Regression, Logistic
Statistical Analysis 4: Comparison: Ankylosing Spondylitis; Remission and participant age; Test type: Superiority or Other; p = 0.0001, Regression, Logistic
Statistical Analysis 5: Comparison: Ankylosing Spondylitis; Remission and positive tuberculosis screening at Visit 0; Test type: Superiority or Other; p = 0.0734, Regression, Logistic
Statistical Analysis 6: Comparison: Ankylosing Spondylitis; Remission and male gender; Test type: Superiority or Other; p = 0.0438, Regression, Logistic
Statistical Analysis 7: Comparison: Ankylosing Spondylitis; Remission and BASDAI score at Visit 0; Test type: Superiority or Other; p = 0.5030, Regression, Logistic

8. Secondary Outcome: Mean Change in Health Assessment Questionnaire Disability Index (HAQ-DI) Score (in Case of Peripheral Symptoms) or Bath Ankylosing Spondylitis Functional Index (BASFI) Score (in Case of Axial Symptoms) in Participants With Ankylosing Spondylitis
Description: HAQ-DI consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, with a higher score representing a high-dependency disability. The minimal clinically important difference defined for the HAQ-DI is ≥0.22. HAQ-DI remission, indicating normal physical function, is defined as HAQ-DI < 0.5. The BASFI is a set of 10 questions designed to determine the degree of functional limitation in those with AS. A visual analogue scale (with 0 being "easy" and 10 "impossible") is used. The BASFI score ranges from 0 to 10 and is derived as the mean of the single items. A higher score indicates a higher impairment of functioning.
Time Frame: Baseline (Visit 0) to 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 346
Units on a scale
  Mean change in HAQ-DI, n=30 | -0.9 (0.6)
  Mean change in BASFI, n=346 | -4.1 (2.5)

9. Secondary Outcome: Mean Frequency of Extra-articular Manifestations (EAMs)
Description: Extra-articular manifestations (EAMs) are symptoms and diseases that occur in parts of the body other than joints. The number of EAMs was determined at each study visit. These included the presence of enthesitis (inflammation of ligaments and/or tendons at the site of insertion into bones), uveitis (inflammation of the middle layer of the eye), psoriasis (a skin condition that causes itchy or sore patches of thick, red skin with silvery scales), and Inflammatory bowel disease (Crohn's disease or ulcerative colitis).
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants who received adalimumab treatment
Measure: Mean (Standard Deviation); unit: Mean EAMs per participant
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 403 | 151
Mean EAMs per participant
  Baseline (Visit 0), n=403, 151 | 0.5 (0.6) | 1.1 (0.6)
  Visit 1 , n=400, 150 | 0.2 (0.4) | 0.6 (0.6)
  Visit 2, n=357, 137 | 0.1 (0.3) | 0.5 (0.6)
  Visit 3, n=339, 124 | 0.1 (0.3) | 0.5 (0.5)
  Visit 4, n=324, 124 | 0.1 (0.3) | 0.5 (0.5)
  Visit 4-LOCF, n=401, 151 | 0.1 (0.3) | 0.5 (0.5)

10. Secondary Outcome: Duration of Treatment With Adalimumab
Description: The duration of treatment with adalimumab was calculated separately for participants who discontinued the medication during the study and for those who did not.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants who received adalimumab treatment
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 381 | 140
Months
  No discontinuation of treatment, n=315, 117 | 11.8 (1.2) | 11.6 (1.1)
  Discontinuation of treatment, n=66, 23 | 4.8 (3.0) | 5.0 (3.2)

11. Secondary Outcome: Percentage of Participants Whose Co-medication With Nonsteroidal Anti-inflammatory Drugs (NSAIDs) Was Stopped During the Study
Description: Participants were surveyed at each study visit for their use of NSAID medication.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants who were receiving NSAID medication at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 265 | 39
Percentage of participants | 96.6 | 94.9

12. Secondary Outcome: Mean Change in Individual Components of the Work Productivity and Activity Impairment Specific Health Problem Questionnaire in Participants With Ankylosing Spondylitis
Description: Work Productivity and Activity Impairment (WPAI) Questionnaire is a quantitative assessment of the amount of absenteeism, presenteeism, total work productivity impairment, and total activity impairment attributable to a specific health problem (WPAI-SHP), expressed as a percentage. Participants were queried regarding their current employment status, hours missed from work because of problems associated with their AS, hours missed from work because of any other reason, number of hours worked, how much AS affected work productivity (0=AS had no effect,10= AS completely prevented me from working), and how much AS affected ability to do regular daily activities, other than work at a job (0= AS had no effect, 10= AS completely prevented me from doing my daily activities) in the past 7 days.
Time Frame: Baseline (Visit 0) to 12 months
Population: For presenteeism, absenteeism, and total work productivity impairment endpoints: participants with ankylosing spondylitis who were employed at the time of the documentation. For the total activity impairment endpoint: participants with ankylosing spondylitis who received adalimumab treatment.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 342
Percentage change
  Mean change in absenteeism, n=170 | -9.7 (24.4)
  Mean change in presenteeism, n=160 | -37.3 (28.0)
  Mean change in work productivity impairment, n=160 | -38.6 (28.8)
  Mean change in total activity impairment, n=342 | -36.5 (26.7)

13. Secondary Outcome: Change in the Percentage of Ankylosing Spondylitis Participants Who Have Paid Work
Description: Working status (Working full-time, working part-time, working at home, unemployed but seeking work, work disabled, retired, student) was documented at each study visit.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with ankylosing spondylitis who received adalimumab treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 403
Percentage of participants
  Working at Baseline (Visit 0), n=403 | 56.6
  Working at last visit- valid data, n=351 | 56.1

14. Secondary Outcome: Mean Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score (in Case of Axial Symptoms) and/or Disease Activity Score/28 Joints (DAS28) (in Case of Peripheral Symptoms) in Participants With Psoriatic Arthritis
Description: as for outcome 4
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with psoriatic arthritis with peripheral symptoms (DAS28 > 5.1 at baseline) and/or active axial symptoms (a baseline value of BASDAI > 4)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 61
Units on a scale
  Mean change in BASDAI score, n=52 | -4.2 (2.4)
  Mean change in DAS28 score, n=61 | -2.4 (1.3)

15. Secondary Outcome: Correlation Between Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Ankylosing Spondylitis Disease Activity Score (ASDAS) in Participants With Psoriatic Arthritis
Description: BASDAI score (ranging from 0 to 10) was calculated using a questionnaire. Participants marked responses on a 10 cm visual analog scale ranging from 0 (none) to 10 (very severe) regarding fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. A positive response was defined as a 50% or more decrease in the BASDAI score at 12 months as compared to baseline. ASDAS score consists of a self-administered questionnaire plus an objective laboratory evaluation. The questionnaire covers disease activity, back pain, duration of morning stiffness and peripheral pain/swelling assessed on a visual analogue scale (from 0 to 10 cm) or on a numerical rating scale (from 0 to 10). The laboratory parameter is a measurement of C-reactive protein (mg/L) or erythrocyte sedimentation rate (mm/h). Spearman's rank correlation coefficient (CC) was calculated for BASDAI vs. ASDAS(subscript)CRP(subscript) and BASDAI vs. ASDAS(subscript)ESR(subscript).
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with psoriatic arthritis and active axial symptoms (a baseline value of BASDAI > 4)
Measure: Number; unit: Correlation coefficient
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 51
Correlation coefficient
  Correlation BASDAI and ASDAS-CRP, n=45 | 0.75
  Correlation BASDAI and ASDAS-ESR, n=51 | 0.84

16. Secondary Outcome: Predictors of Maintained Treatment Response and Remission in Participants With Psoriatic Arthritis
Description: as for outcome 7
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with psoriatic arthritis and active axial symptoms (a baseline value of BASDAI > 4)
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 52
Odds Ratio
  Treatment response (Enthesitis at Visit 0) | 0.23 [0.05 to 1.05]
  Treatment response (BASDAI score at Visit 0) | 1.35 [0.88 to 2.08]
  Remission (Psoriasis at Visit 0) | 0.21 [0.04 to 1.16]
  Remission (BASDAI score at Visit 0) | 0.87 [0.58 to 1.31]
Statistical Analysis 1: Comparison: Psoriatic Arthritis; Treatment response and presence of enthesitis at Visit 0; Test type: Superiority or Other; p = 0.0576, Regression, Logistic
Statistical Analysis 2: Comparison: Psoriatic Arthritis; Treatment response and BASDAI score at Visit 0; Test type: Superiority or Other; p = 0.1739, Regression, Logistic
Statistical Analysis 3: Comparison: Psoriatic Arthritis; Remission and Psoriasis at Visit 0; Test type: Superiority or Other; p = 0.0733, Regression, Logistic
Statistical Analysis 4: Comparison: Psoriatic Arthritis; Remission and BASDAI at Visit 0; Test type: Superiority or Other; p = 0.5000, Regression, Logistic

17. Secondary Outcome: Mean Change in Health Assessment Questionnaire Disability Index ( HAQ-DI) Score (in Case of Peripheral Symptoms) or Bath Ankylosing Spondylitis Functional Index (BASFI) Score (in Case of Axial Symptoms) in Participants With Psoriatic Arthritis
Description: as for outcome 8
Time Frame: Baseline (Visit 0) to 12 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 88
Units on a scale
  Mean change in HAQ-DI, n=88 | -0.7 (0.6)
  Mean change in BASFI, n=47 | -3.8 (2.8)

18. Secondary Outcome: Mean Change in Individual Components of the Work Productivity and Activity Impairment Specific Health Problem Questionnaire in Participants With Psoriatic Arthritis
Description: The Work Productivity and Activity Impairment (WPAI) Questionnaire is a quantitative assessment of the amount of absenteeism, presenteeism, total work productivity impairment, and total activity impairment attributable to a specific health problem (WPAI-SHP), expressed as a percentage. Participants were queried regarding their current employment status, hours missed from work because of problems associated with their PsA, hours missed from work because of any other reason, number of hours worked, how much PsA affected work productivity (0= PsA had no effect,10= PsA completely prevented me from working), and how much PsA affected ability to do regular daily activities, other than work at a job (0= PsA had no effect, 10= PsA completely prevented me from doing my daily activities) in the past 7 days.
Time Frame: Baseline (Visit 0) to 12 months
Population: For presenteeism, absenteeism, and total work productivity impairment endpoints: participants with psoriatic arthritis who were employed at the time of the documentation. For the total activity impairment endpoint: participants with psoriatic arthritis who received adalimumab treatment.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 119
Percentage change
  Mean change in absenteeism, n=57 | -6.0 (29.0)
  Mean change in presenteeism, n=54 | -32.8 (24.9)
  Mean change in work productivity impairment, n=54 | -33.6 (25.4)
  Mean change in total activity impairment, n=119 | -34.7 (25.7)

19. Primary Outcome: Percentage of Participants With Peripheral Symptoms in Remission
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Remission was defined as DAS28 ≤2.6 at 12 months.
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with peripheral symptoms (DAS28 > 5.1 at baseline)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis | Psoriatic Arthritis
Number analyzed (Participants) | 18 | 61
Percentage of participants | 11.1 [1.4 to 34.7] | 14.8 [7.0 to 26.2]

20. Secondary Outcome: Change in the Percentage of Psoriatic Arthritis Participants Who Have Paid Work
Description: as for outcome 13
Time Frame: Baseline (Visit 0) to 12 months
Population: Participants with psoriatic arthritis who received adalimumab treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 151
Percentage of participants
  Working at Baseline (Visit 0), n=151 | 55.6
  Working at last visit- valid data, n=140 | 54.3

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of adalimumab administration until the completion of the study, up to 52 weeks.
Description: In case of premature discontinuation, participants were followed for 70 days (5 half-lives) following the intake of the last dose of adalimumab.
Groups:
- Overall Study Population: Participants who received adalimumab treatment
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 26/555
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Population (N=555)
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral mucosal blistering (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Feeling abnormal (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site rash (General disorders) | 1
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Erysipelas (Infections and infestations) | 1
Lymphadenitis bacterial (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Morphoea (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Hip surgery (Surgical and medical procedures) | 1
Lymphadenectomy (Surgical and medical procedures) | 1
Phlebectomy (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.